CLINICAL TRIAL: NCT05744830
Title: The Effect of a Single Implant Retained Removable Complete Overdenture in the Mandible on Hearing Ability of Edentulous Patients- Randomised Controlled Trial
Brief Title: The Effect of a Removable Complete Denture Over One Implant in the Lower Jaw on Hearing Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: Al Mouwasat Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Prosth-01-2023
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hearing
Keywords: Bone Conduction; Pure Tone Audiometry(PTA); Hearing ability; Single implant
MeSH Terms: interventions — Denture, Overlay; Denture, Complete

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blinding, the physician who does the audiogram
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overdenture (Experimental): Each patient in this group will receive a single implant overdenture.
  Interventions: Other: Overdenture
- Complete Denture (Experimental): Each patient in this group will receive a removable complete denture without implants.
  Interventions: Other: Complete Denture

INTERVENTIONS:
Other: Overdenture — 15 patients will receive removable complete dentures, then a single implant is placed in the midline of the mandible, then loaded with the denture.
  Arms: Overdenture
Other: Complete Denture — 15 patients will only receive removable complete dentures
  Arms: Complete Denture

SUMMARY:
The effect of a removable complete denture and the insertion of one implant in the lower jaw and the loading of this implant on the hearing ability of patients will be studied, so the hearing ability will be measured by using the PTA test for 30 patients in the age of 50-65 years old. The hearing ability measurement will be done in 4 different periods of time. Before and after using the denture, before and after the implant insertion, and after loading the implant with the same complete denture. The implant surgery will be done in two phases: the first is to insert the implant in the bone and cover it by suturing until it integrates with the bone after 3 months, the second is to start the process of loading the implant with the denture.

DETAILED DESCRIPTION:
Tanaka et al mentioned in their study that in accordance to the WHO, about one third of the people older than 65 years old is somehow affected by hearing loss. Although hearing loss is not a life-threatening condition but it is related to medical and psychological problems such as depression and social isolation. Reduction in the occlusal vertical dimension is considered one of the factors that cause a decline in hearing ability. A study of Shreedhar et al found that there is improvement in hearing ability between loading two implants in the canine regions in the mandible with a removable complete overdenture and after one month of the loading. In their study, the hearing threshold improved from 40 to 25 decibel and the improvement is associated with transmission of vibrations from the oral cavity through the bone. Implants in the mandible has been associated with improvement in hearing although the mandible is not in direct contact with the skull, and Ozer et al study found that the hearing acuity through the bone was not different between the upper and lower jaw. In Tanaka et al study teeth loss was associated with the increased prevalence of hearing loss. King et al found important improvement in previously existed hearing loss after the replacement of missing teeth with a removable complete overdenture. Furthermore, Schell et al study found that hearing acuity was worse in the edentulous patients group than the other groups, which suggests a relation between hearing loss and the dentate status. A similar study of Peeters et al mentioned that the discrepancy between patients who had complete dentures and patients who had loss in the occlusal vertical dimension strengthen the hypothesis that there is an association between hearing loss and the occlusal vertical dimension. As for the single implant retained complete overdenture, there has been several studies, which are mentioned in carl's Misch book that found this treatment to be valid, especially for patients who suffer from removable dentures and have problems in mastication.

The available evidence on the relationship between dentate status and hearing loss is limited, so understanding this relationship could help prevent or delay the occurrence of hearing loss. The possibility of suggesting implant placement and loading the implant with a removable complete overdenture as a way to improve bone-conducted hearing in edentulous patients will be studied.

In this study, we are going to measure the hearing ability of edentulous patients 4 times: First, before using the complete denture. Second, after using it for one month and before placing the implant. Third, 10 days after placing the implant in the midline of the mandibular jaw. Fourth, after 1 month of loading the implant with the removable complete overdenture. The null hypothesis is that there is no statistically important difference in hearing thresholds by bone conduction between the studied periods of time. This study will be done on 30 patients and a written consent will be taken. The hearing ability test will be done in Al-Mowasat hospital after the examination of the patient by an otolaryngologist before the first hearing test. The hearing ability test is called Pure Tone Audiometry or PTA.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-65 years old.
* No previous experience in removable complete dentures.
* Enough bone in the midline of the mandibular jaw that permits the placement of a single implant no less than 10 mm in length and 3.4 mm in width.
* Hearing threshold of the patient between 40-70 decibel.
* The ability of the patient to fill out the questionnaire and commit to follow up sessions.

Exclusion Criteria:

Having one of the variables that are connected with hearing loss, which are:

* usage of hearing aids.
* Uncontrolled diabetes.
* Uncontrolled hypertension.
* Balance problems.

In addition to risk factors that are associated with hearing loss, which are:

* stroke
* kidney disease

In addition to contraindications for implant surgery, which are:

1. definitive contraindications: Recent myocardial infarction, valve replacements, cardiovascular diseases ,and presence of immunodeficiency, bleeding problems, drug abuse, and psychological disease.
2. Relative contraindications:

Osteoporosis, heavy smoking, uncontrolled diabetes, hypothyroidism.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Hearing ability of edentulous patients | hearing ability will be measured 3 days before and 1 month after using the removable complete denture.
  Hearing ability is expressed in the present study as hearing threshold (HT) measured by pure tone audiometry (PTA). PTA is performed by producing auditory stimuli from headphones strating from 30 decibels (dB). A gradual increase by 15dB is implemented until HT is reached. HT value is recorded when the participant hears the lowest tone and raises his/her hand.

CONTACTS AND LOCATIONS:
Overall Officials: Lujain Jadaan, DDS, Principal Investigator — MSc student, Department of Prosthodotics, University of Damascus Dental School, Damascus; Ammar Almustafa, DDS MSc PhD, Study Director — Assistant Professor, Department of Prosthodotics, University of Damascus Dental School, Damascus; Samer Mohsen, MD MSc PhD, Study Director — Assistant Professor, Department of Audiology, Faculty of Medicine, Damascus University
Locations (1):
- Department of removable prosthodontics, University of Damascus Dental School, Damascus, Dimashq, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krennmair G, Ulm C. The symphyseal single-tooth implant for anchorage of a mandibular complete denture in geriatric patients: a clinical report. Int J Oral Maxillofac Implants. 2001 Jan-Feb;16(1):98-104. PMID 11280368
- [Background] Lawrence HP, Garcia RI, Essick GK, Hawkins R, Krall EA, Spiro A 3rd, Vokonas PS, Kong L, King T, Koch GG. A longitudinal study of the association between tooth loss and age-related hearing loss. Spec Care Dentist. 2001 Jul-Aug;21(4):129-40. doi: 10.1111/j.1754-4505.2001.tb00242.x. PMID 11669061
- [Background] Liddelow G, Henry P. The immediately loaded single implant-retained mandibular overdenture: a 36-month prospective study. Int J Prosthodont. 2010 Jan-Feb;23(1):13-21. PMID 20234886
- [Background] Nagasaka H, Matsukubo T, Takaesu Y, Kobayashi Y, Sato T, Ishikawa T. Changes and equalization in hearing level induced by dental treatment and instruction in bilaterally equalized chewing: a clinical report. Bull Tokyo Dent Coll. 2002 Nov;43(4):243-50. doi: 10.2209/tdcpublication.43.243. PMID 12687730
- [Background] Peeters J, Naert I, Carette E, Manders E, Jacobs R. A potential link between oral status and hearing impairment: preliminary observations. J Oral Rehabil. 2004 Apr;31(4):306-10. doi: 10.1046/j.1365-2842.2003.01252.x. PMID 15089934
- [Background] Shreedhar S, Raza FB, Vaidyanathan AK, Veeravalli PT. Effect of an implant-retained complete overdenture on the hearing ability of edentulous patients: A clinical pilot study. J Prosthet Dent. 2021 Apr;125(4):628-635. doi: 10.1016/j.prosdent.2020.02.015. Epub 2020 Apr 26. PMID 32345511
- [Derived] Jadaan L, Mohsen S, Almustafa A. Hearing of Edentulous Patients With a Single Implant-Retained Removable Complete Overdenture: A Case Series. Spec Care Dentist. 2026 Jan-Feb;46(1):e70138. doi: 10.1111/scd.70138. PMID 41521677